CLINICAL TRIAL: NCT04662814
Title: the Efficacy of Extracorporeal Shock Wave Therapy for Primary Dysmenorrhea
Brief Title: Extracorporeal Shock Wave Therapy for Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Collaborators: Ghada ebrahim El Refaye -Faculty of Physical Therapy, Cairo University, Egypt (Unknown); Sohier Mahmmoud El Koseiry- Faculty of Physical Therapy, Cairo University, Egypt (Unknown)
Responsible Party: Principal Investigator, shaimaa Mohamed hamed, principle investigator, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mtiu
Record Dates: First submitted 2020-11-22; First posted 2020-12-10 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Diet Therapy

STUDY DESIGN:
Intervention Model Description: group A: shockwave therapy and dietary modification group B: dietary modification
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shock wave (Experimental): shock wave for primary dysmenorrhea for study group along side to dietary modification
  Interventions: Other: shock wave therapy; Other: dietary modification
- dietary modification (Active Comparator): dietary modification for primary dysmenorrhea for control group
  Interventions: Other: dietary modification

INTERVENTIONS:
Other: shock wave therapy — Intervention group is by shock wave therapy. A radial shock wave device (EME, ITALY) was used. for 4 sessions (one session before the expected day of period and session per day for day1 , day 2 and day 3 of each menstrual cycle) for three successive periods.
  Arms: shock wave
Other: dietary modification — Participants will receive dietary modification for three consecutive months dietary modification will be low caffeine and high water and liquids intake and reduce the uptake of fast food, should be followed for 3 months

SUMMARY:
purpose of this study to investigate the effect of Extracorporeal shock wave therapy on pain and prostaglandin level in patient with primary dysmenorrhea

DETAILED DESCRIPTION:
This randomized controlled trial is to determine the effect of shock wave therapy in the treatment of primary dysmenorrhea.

females are randomly assigned into 2 groups: group A SWT treatment plus dietary modification during PD (n=25） GROUP B:dietary modification only (n=25）;

Participants in group B will receive dietary modification for three successive months

The numerical rating scale (NRS) and prostaglandin blood level will be recorded and evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ages ranged between18 - 25 years old.
2. body mass index (BMI) will not exceed 30kg/m2.
3. females will be diagnosed by the physician as primary dysmenorrhea.

Exclusion Criteria:

1. Secondary dysmenorrhea .
2. Mental health problem such as depression and anxiety.
3. Irregular periods

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
numerical rating scale | 3 months
  Numeric rating scale will be 10 cm digital line with 0 (zero) representing feeling no pain and 10 representing feeling the worst pain, was used to assess the severity of the pain before and after treatment for all females in both groups (A&B).
  measurement will done twice first one at baseline(will be considered as pre treatment measure) and 2nd on e at 3rd menstrual cycle ( will be considered as post treatment measure)

SECONDARY OUTCOMES:
prostaglandin | 3months
  5cm plasma concentrations of prostaglandin F2α was taken from all females and was analyzed in the Laboratory index to determine the prostaglandin plasma level
  measurement will done twice before after the treatment program.

CONTACTS AND LOCATIONS:
Locations (1):
- MTI, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT04662814/Prot_ICF_000.pdf